CLINICAL TRIAL: NCT06317987
Title: Addressing Barriers to Care for Substance Use Disorder Pilot Study (Center for Dissemination and Implementation At Stanford, Research Component #3)
Brief Title: Addressing Barriers to Care for Substance Use Disorder Pilot Study
Acronym: ABCSUD Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Stanford University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joseph Glass, Senior Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2068557; P50DA054072 (NIH)
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Drug Use Disorders; Illicit Drug Use; Alcohol-Related Disorders
Keywords: Implementation Science; Care Navigation; Drug Use Disorders; Quality Improvement; Behavioral Health
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Care coordinators were randomized to two parallel groups: usual care (UC; i.e., the comparator group) and usual care plus care navigation (UC + CN; i.e., the experimental group). All care coordinators continued offering substance use resources and treatment options to patients as usual. Clinicians randomized to UC + CN were able to offer and refer patients to a care navigator.
Who Masked: Outcomes Assessor
Masking Description: All study outcomes are extracted from secondary data including electronic health record and healthcare claims databases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care Navigation (pilot) (Experimental): Mental health care coordinators offer and refer patients to a care navigator in addition to offering substance use resources and treatment options as usual.
  Interventions: Behavioral: Care Navigation
- Services as Usual (pilot) (No Intervention): Mental health care coordinators offer substance use resources and treatment options to patients as usual

INTERVENTIONS:
Behavioral: Care Navigation — Care navigation is an intervention that seeks to help patients follow up on substance use treatment plans that are established by care coordinators in the health system by reducing barriers to accessing treatment. This includes advocating for patients to reduce disparities based on language, income or geographical barriers, and cultural preferences (i.e., linkage to available services); and using motivational enhancement techniques to help patients maintain their motivation to obtain substance use treatment while working through these barriers (i.e., motivational intervention). Thus, the care navigator's role is to take the care plan developed between the patient and the mental health care coordinator forward and connect the patient to available services and provide motivational enhancement techniques to help direct the patient toward completion of the care plan.
  Arms: Care Navigation (pilot)

SUMMARY:
The Addressing Barriers to Care for Substance Use Disorder Pilot (ABC-SUD Pilot) was a randomized pilot study that preceded a larger trial. The ABC-SUD Pilot was a parallel group, cluster-randomized pilot feasibility trial, with clinicians (care coordinators) as the unit of randomization.

This study was conducted in a mental health treatment access center within the Washington region of Kaiser Permanente. As part of usual care, patients contacted the mental health access center to speak to a "care coordinator" to obtain contact information for potential venues to obtain treatment for substance use disorder.

The experimental intervention, Care Navigation, was evaluated for its potential to increase the utilization of substance use disorder treatment among patients who contacted the mental health treatment access center. The investigators note that Care Navigation was delivered by study "care navigators", who were distinct from the health system's care coordinators.

DETAILED DESCRIPTION:
The ABC-SUD Pilot was conducted to evaluate feasibility of conducting a larger trial. Specific goals were to a) confirm patient eligibility criteria, b) confirm selection of the primary and secondary outcomes and the approach to measuring them using electronic health record data, c) confirm the feasibility and acceptability of randomization procedures, d) evaluate the feasibility of care navigation protocol delivery by care coordinators, e) evaluate feasibility of electronic health record templates to assist care coordinators when referring patients to care navigators. This pilot also helped refine study implementation needs and statistical analysis plans for the trial.

The pilot's recruitment goal was to offer care navigation to patients until a total of 10 patients agreed to care navigation. The investigators conducted post-intervention quality improvement interviews with several enrolled patients to obtain feedback on intervention design to inform changes.

To recruit care coordinators for the pilot, mental health treatment access center managers identified 4 care coordinators who volunteered to participate in piloting the care navigator intervention.

To maximize the study sample for the larger trial, the pilot evaluated the feasibility of employing a "vanguard" randomization approach, which is a type of stratified randomization in which pilot (or vanguard) care coordinators are pre-randomized to begin piloting the intervention but then retain their randomization status for the subsequent trial. When using the vanguard method, the patient eligibility for the pilot period and trial period are distinct.

Clinicians (care coordinators) were eligible if they conduct video or phone-based assessment and treatment planning visits in the mental health treatment access center, had been employed for at least 1 month, had completed trainings related to their clinical role in the health system, were scheduled to conduct at least 3 assessments per day, and consented to participate in the study.

Over the course of the pilot, we changed patient eligibility criteria. During the first period of the pilot (07/09/2024 - 09/15/2024), the sample of patients eligible for the pilot analyses included individuals with a visit to an enrolled care coordinator who were ≥ 18 years of age and have a SUD assessment and treatment planning visit with a care coordinator. During the second period of the pilot (09/16/2024 - 11/27/2024), the sample of patients eligible for the pilot analyses included individuals with a visit to an enrolled care coordinator during the patient eligibility period who were ≥ 18 years of age, engaged in substance use, and had a mental health assessment and treatment planning visit with a care coordinator. We switched the eligibility criteria to allow us to determine the feasibility and appropriateness of offering care navigation to people with substance use who were seeking mental health treatment (instead of substance use treatment).

Analyses follow an intent-to-treat principle whereby care coordinators are analyzed according to the intervention arm to which they were randomized regardless of the subsequent sequence of events. The patient eligibility period was defined as the period in which patients become eligible for the study (i.e., for inclusion in the analytic sample). This period is anticipated to start within 2 weeks of the clinician's randomization date (to allow for sufficient time for intervention coordinators to be trained). The investigators anticipated that approximately 40 patients would comprise the analytic sample.

ELIGIBILITY:
Clinician (Care Coordinator) Inclusion Criteria:

* Conducts video or phone-based assessment and treatment planning visits in the mental health treatment access center
* Has been employed for at least 1 month and has completed trainings related to their clinical role in the health system
* Scheduled to conduct at least 3 assessments per day
* Has consented to participate in the study.

Clinician Exclusion Criteria:

- None

Patient Inclusion Criteria (eligibility for analyses):

* Visits an enrolled care coordinator during the patient eligibility period
* ≥ 18 years of age at the time of the visit
* Has an assessment and treatment planning visit for SUD with an enrolled care coordinator (this criterion was applied during the first period of the pilot, 7/9/2024-9/15/2024)
* Has evidence of substance use as determined by the care coordinator (this criterion was applied during the second period of the pilot, 9/16/2024-11/27/2024)
* Has an assessment and treatment planning visit for mental health treatment with an enrolled care coordinator (this criterion was applied during the second period of the pilot, 9/16/2024-11/27/2024)

Patient Exclusion Criteria:

* Patients who have requested through the health system to opt out of research contact or chart review
* Patients who are not enrolled in Kaiser Permanente or Medicaid insurance (anticipated incomplete capture of covariate and/or outcome information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patient interest in care navigation | From pilot study launch to end of accrual (anticipated 16 weeks; see recruitment goals above)
  Proportion of patients who agree to a care coordinator's offer to be contacted by a care navigator

SECONDARY OUTCOMES:
Feasibility of patient consent procedures | From study launch to end of accrual (anticipated 16 weeks; see recruitment goals above)
  Proportion of patients who consent to the study among those who agree to be contacted by a care navigator

OTHER OUTCOMES:
SUD treatment - 30 days | Time Frame: From patient's clinical assessment appointment to 30 days later
  Proportion of patients who utilize treatment within 30 days
SUD treatment - 60 days | Time Frame: From patient's clinical assessment appointment to 60 days later
  Proportion of patients who utilize treatment within 60 days
SUD treatment - 90 days | Time Frame: From patient's clinical assessment appointment to 90 days later
  Proportion of patients who utilize treatment within 90 days
SUD treatment visits - 30 days | Time Frame: From patient's clinical assessment appointment to 30 days later
  Number of SUD treatment visits within 30 days
SUD treatment visits - 60 days | Time Frame: From patient's clinical assessment appointment to 60 days later
  Number of SUD treatment visits within 60 days
SUD treatment visits - 90 days | Time Frame: From patient's clinical assessment appointment to 90 days later
  Number of SUD treatment visits within 90 days
Days until SUD treatment utilization from clinical assessment appointment | From patient's clinical assessment appointment to up to 90 days later
  Time-to-event measure of SUD treatment utilization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Glass, PhD, MSW, Principal Investigator — Chestnut Health Systems Inc
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
This study protocol is embedded within a Center of Excellence funded by the National Institute on Drug Abuse. In coordination with other center project components, the study protocol will be submitted for publication to either an addiction or implementation science journal. Additional data (analytic code) can be requested from the Principal Investigator. Participant data will be shared with the prime site as allowed. Analysis files will be constructed from the electronic data and aggregated. No names, addresses, telephone numbers, email addresses, medical record numbers, etc. will be retained in the aggregated files.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: To be determined
Access Criteria: Access criteria will be determined by Kaiser Permanente and Stanford University